CLINICAL TRIAL: NCT05049629
Title: Effect of Chitosan-N-Acetylcysteine (Lacrimera®) on IOL-power Prior to Cataract Surgery: a Pilot Study
Brief Title: Effect of Chitosan-N-Acetylcysteine on IOL-power Prior to Cataract Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Medical device expired
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Lacrimera Biometry
Record Dates: First submitted 2021-09-01; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Intervention Model Description: After enrolment into the study three study visits will be scheduled. The selection of the study eye will be randomized using www.randomizer.org. The contralateral eye serves as the control eye. After the baseline examination and the follow-up examination one hour later, patients will be released with a prescription of one drop of Lacrimera® into the study eye per day in the evening and with one drop of single-use preservative-free hyaluronic acid containing eye drops (Hylo-Vision® sine) into the control eye three times a day for 14 consecutive days.
Masking Description: All study-related measurements will be performed by a masked observer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye 1 (Experimental): The contralateral eye serves as the control eye. After the baseline examination and the follow-up examination one hour later, patients will be released with a prescription of one drop of Lacrimera® into the study eye per day in the evening and with one drop of single-use preservative-free hyaluronic acid containing eye drops (Hylo-Vision® sine) into the control eye three times a day for 14 consecutive days.
  Interventions: Device: Lacrimera
- Eye 2 (Active Comparator): The contralateral eye serves as the control eye. After the baseline examination and the follow-up examination one hour later, patients will be released with a prescription of one drop of Lacrimera® into the study eye per day in the evening and with one drop of single-use preservative-free hyaluronic acid containing eye drops (Hylo-Vision® sine) into the control eye three times a day for 14 consecutive days.
  Interventions: Device: Hylo-Vision

INTERVENTIONS:
Device: Lacrimera — A new preservative-free formulation of eye drops consists of a novel biopolymer, chitosan-N-acetylcysteine (C-NAC; Lacrimera®, Croma-Pharma GmbH, Leobendorf, Austria), which electrostatically binds to the mucine layer of the tear film forming a glycocalyx-like structure.
  Arms: Eye 1
Device: Hylo-Vision — Preservative-free, Hyaluronic-acid containing eyedrops (Hylo-Vision® sine)
  Arms: Eye 2

SUMMARY:
Aim of this study is to evaluate the effect of treatment with Lacrimera® on calculated IOL power prior to cataract surgery and on the stability of ocular surface parameters compared to preservative-free, Hyaluronic-acid containing eyedrops (Hylo-Vision® sine).

DETAILED DESCRIPTION:
The present study seeks to investigate the effect of treatment with Lacrimera® on the calculated IOL power prior to cataract surgery and on the stability of ocular surface parameters compared to preservative-free, Hyaluronic-acid containing eyedrops (Hylo-Vision® sine).

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Corneal staining (marked to severe; NEI grading scale >=10)

Exclusion Criteria:

* Usage of eye drops other than lubricants (e.g. antibiotics, steroids, cyclosporin-A)
* Usage of systemic antibiotic therapy 7
* Any pathology of the ocular surface except dry eye disease (e.g. corneal scarring, cornea ectasia)
* Ocular surgery within prior 3 months
* Preceding refractive surgery (e.g. LASIK)
* Ocular injury within prior 3 months
* Ocular herpes of eye or eyelid within prior 3 months
* Active ocular infection
* Active ocular inflammation or history of chronic, recurrent ocular inflammation within prior 3 months
* Eyelid abnormalities that affect lid function
* Ocular surface abnormality that may compromise corneal integrity
* Pregnancy and nursing women (in women of childbearing age a pregnancy test will be performed before inclusion into the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Spherical and toric IOL power | 1 hour
  Spherical and toric IOL power selected at baseline
Spherical and toric IOL power | 2 weeks
  Spherical and toric IOL power selected at the 2 weeks visit
Difference in spherical and toric IOL power | 2 weeks
  Difference in spherical and toric IOL power between baseline and the 2 weeks visit

SECONDARY OUTCOMES:
Reproducibility of biometry readings | 2 weeks +/- 2 days
  Reproducibility of biometry readings at each study visit (Baseline, 1 hour after Baseline, after 1 week, after 2 weeks)
  * Axial length
  * Keratometry readings (K1, K2)
Change of dry eye parameters | 2 weeks +/- 2 days
  Change of dry eye parameters between baseline and 2 weeks
  * BUT (fluorescein and non-invasive BUT)
  * NEI grading score
Difference between study and control eye | 2 weeks +/- 2 days
  Difference between study and control eye (baseline and 2 weeks)
  * BUT (fluorescein and non-invasive BUT)
  * NEI grading score

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, PrimUnivPrDr, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No